CLINICAL TRIAL: NCT04475094
Title: Impact of Coronary Artery Stenting on Quantitative Myocardial Blood Flow and Health Status
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiovascular Imaging Technologies (Industry)
Responsible Party: Principal Investigator, Timothy M. Bateman, MD, Medical Director, Cardiovascular Imaging Technologies
Other Study IDs: 19-080
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial Blood Flow
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rubidium-82

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COHORT: All patients will have had a clinically-indicated PET revealing at least one reversible perfusion defect followed by a research-indicated cardiac PET study between 3 and 8 weeks post-successful coronary artery stenting.
  Interventions: Drug: Rubidium-82; Behavioral: Seattle Angina Questionnaire-7; Behavioral: Rose Dyspnea Scale

INTERVENTIONS:
Drug: Rubidium-82 — Consented subjects will undergo a rest/regadenoson stress myocardial perfusion PET study.
  Other Names: Myocardial Perfusion PET
Behavioral: Seattle Angina Questionnaire-7 — Consented subjects will complete a SAQ-7.
Behavioral: Rose Dyspnea Scale — Consented subjects will complete a RDS.

SUMMARY:
We propose to perform PET MPI studies in patients before and after stenting to evaluate changes (or lack thereof) in MBFR and how that is associated with changes (or lack thereof) in symptoms, functional status and quality of life. This will help to understand the role of MBFR in patient selection for coronary angiography and stenting.

DETAILED DESCRIPTION:
Myocardial perfusion imaging (MPI) has a well-established role in diagnosis, risk stratification and prognostication in patients with suspected or known coronary artery disease (CAD)(1,2). As the current health-care landscape moves towards rewarding value, there is an increased urgency for determining the role of imaging tests in improving patient-centered outcomes (3-5). Traditionally, the cardiac imaging community has focused on studying "hard outcomes" such as cardiac morbidity and mortality, with relatively little attention on patient-centered health status outcomes (e.g. symptoms, function and quality of life).

While Single Photon Emission Computed Tomography (SPECT) has been a myocardial perfusion imaging (MPI) mainstay for decades, use of Positron Emission Tomography (PET) MPI has been increasing as it offers superior spatial resolution, lower radiation exposure, higher diagnostic accuracy, shorter acquisition times and quantification of myocardial blood flow reserve (MBFR) (6-9). MBFR integrates the hemodynamic effects of microvascular dysfunction, diffuse atherosclerotic disease and epicardial stenosis on myocardial tissue perfusion, and as such is more likely to correlate with patient's anginal symptoms, functional status and quality of life (10,11). MBFR measured by PET MPI has been shown to provide independent and incremental prognostic value for major adverse cardiac events beyond perfusion defect analysis, but has not been evaluated for its association with symptoms, function and quality of life (although in a post-hoc analysis of 171 patients with known CAD undergoing PET MPI enrolled in the ASPIRE study at our center, higher MBFR was significantly associated with lower anginal burden as measured by the Seattle Angina Questionnaire (SAQ; unpublished data, being presented at ASNC 2018)) (8,10,12-15). Among 329 patients, Taqueti et al demonstrated that patients with low global MBFR were less likely to require subsequent heart failure hospitalizations and cardiac deaths if treated with early revascularization with bypass surgery, but not percutaneous coronary intervention (PCI), as compared with medical management; however the low number of events and the small sample size were major limiting factors (10). More recently, among 12,594 patients undergoing PET MPI, we demonstrated that MBFR <1.8 may help identify patients with a survival benefit from early revascularization within 90 days of the index MPI test. (unpublished data, being presented at AHA 2018). In a sub-study of the PACIFIC study, Driessen et al showed strong correlation of change in MBFR post revascularization with change in FFR; providing further support for non-invasively measured MBFR as a potential measure to target intervention, similar to FFR, which needs invasive measurement on coronary angiography (16).

To further elucidate the mechanism of action by which MBFR could be used to target management for ischemic heart disease, we propose a study of serial PET MPI in 75 patients undergoing coronary stenting to evaluate the association of changes in MBFR with changes in patients' health status. About a quarter to half of stable CAD patients treated with PCI continue to have angina and poor quality of life after stenting (17-19) This may be because stenting is only directed at epicardial stenoses, while many patients have concomitant microvascular disease. While there has been some data where serial PET MPI studies have been used to look at changes in perfusion defect sizes and flows with anti-ischemic medications and statins (20-24) it is not known whether these changes are associated with improved outcomes. We propose to perform PET MPI studies in patients before and after stenting to evaluate changes (or lack thereof) in MBFR and how that is associated with changes (or lack thereof) in symptoms, functional status and quality of life. This will help to understand the role of MBFR in patient selection for coronary angiography and stenting.

ELIGIBILITY:
Inclusion Criteria:

1. The index clinically-indicated rest/regadenoson stress myocardial perfusion PET study shows at least one reversible perfusion defect; and
2. The MBFR measurement meets quality control criteria for accuracy; and
3. The patient has completed a baseline SAQ-7 and RDS survey with a SAQ-7 Angina Frequency Score <100 (indicating the occurrence of at least some angina symptoms over the past 4 weeks); and
4. The patient has undergone a successful coronary artery stenting within 60 days after the PET scan without a significant change in clinical condition between the time of baseline PET MPI test and PCI; and 5. The patient agrees to undergo a second PET scan 3-6 weeks after coronary artery stenting and to complete a second SAQ-7 and RDS survey.

Exclusion Criteria:

1. EF <40%
2. Significant aortic stenosis/regurgitation
3. Significant Mitral stenosis/regurgitation)
4. Prior CABG
5. Poor quality base line PET study due one or more technical challenges (e.g. patient motion, imprecise registration of CT and emission data, flows that violate quality criteria, lack of flow augmentation suggestive of an A2A antagonist)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will have had a clinically-indicated PET revealing at least one reversible perfusion defect followed by a research-indicated cardiac PET study between 3 and 8 weeks post-successful coronary artery stenting.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in SAQ-7 Angina Frequency | 3-8 weeks
  The primary study objective is to estimate the association of change from baseline in MBFR with SAQ-7 Angina Frequency scores, adjusting for baseline MBFR, baseline SAQ and other patient factors.
Change in MBFR | 3-8 weeks
  Secondary objective is to estimate the association of change in MBFR with adjusted SAQ-7 Physical Limitation, Quality of Life and Summary scores and Rose Dyspnea Scores (RDS).
Extent of Epicaridal Stenoses | 3-8 weeks
  Exploratory objectives include estimating the association of the extent of epicardial stenoses (vs. microvascular disease) at baseline with post-stent MBFR, SAQ-7 and RDS scores, adjusting for baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luke's Hospital Imaging Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fihn SD, Gardin JM, Abrams J, Berra K, Blankenship JC, Dallas AP, Douglas PS, Foody JM, Gerber TC, Hinderliter AL, King SB 3rd, Kligfield PD, Krumholz HM, Kwong RY, Lim MJ, Linderbaum JA, Mack MJ, Munger MA, Prager RL, Sabik JF, Shaw LJ, Sikkema JD, Smith CR Jr, Smith SC Jr, Spertus JA, Williams SV, Anderson JL; American College of Cardiology Foundation/American Heart Association Task Force. 2012 ACCF/AHA/ACP/AATS/PCNA/SCAI/STS guideline for the diagnosis and management of patients with stable ischemic heart disease: a report of the American College of Cardiology Foundation/American Heart Association task force on practice guidelines, and the American College of Physicians, American Association for Thoracic Surgery, Preventive Cardiovascular Nurses Association, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. Circulation. 2012 Dec 18;126(25):e354-471. doi: 10.1161/CIR.0b013e318277d6a0. Epub 2012 Nov 19. No abstract available. PMID 23166211
- [Background] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Background] Shaw LJ, Blankstein R, Jacobs JE, Leipsic JA, Kwong RY, Taqueti VR, Beanlands RSB, Mieres JH, Flamm SD, Gerber TC, Spertus J, Di Carli MF; American Heart Association Cardiovascular Imaging and Intervention Subcommittee of the Council on Clinical Cardiology; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Cardiovascular Disease in the Young; and Council on Quality of Care and Outcomes Research. Defining Quality in Cardiovascular Imaging: A Scientific Statement From the American Heart Association. Circ Cardiovasc Imaging. 2017 Dec;10(12):e000017. doi: 10.1161/HCI.0000000000000017. PMID 29242239
- [Background] Douglas PS, Cerqueira MD, Berman DS, Chinnaiyan K, Cohen MS, Lundbye JB, Patel RA, Sengupta PP, Soman P, Weissman NJ, Wong TC; ACC Cardiovascular Imaging Council. The Future of Cardiac Imaging: Report of a Think Tank Convened by the American College of Cardiology. JACC Cardiovasc Imaging. 2016 Oct;9(10):1211-1223. doi: 10.1016/j.jcmg.2016.02.027. PMID 27712724
- [Background] Fordyce CB, Douglas PS. Outcomes-Based CV Imaging Research Endpoints and Trial Design: From Pixels to Patient Satisfaction. JACC Cardiovasc Imaging. 2017 Mar;10(3):253-263. doi: 10.1016/j.jcmg.2017.01.010. PMID 28279373
- [Background] Bateman TM, Heller GV, McGhie AI, Friedman JD, Case JA, Bryngelson JR, Hertenstein GK, Moutray KL, Reid K, Cullom SJ. Diagnostic accuracy of rest/stress ECG-gated Rb-82 myocardial perfusion PET: comparison with ECG-gated Tc-99m sestamibi SPECT. J Nucl Cardiol. 2006 Jan-Feb;13(1):24-33. doi: 10.1016/j.nuclcard.2005.12.004. PMID 16464714
- [Background] Danad I, Raijmakers PG, Driessen RS, Leipsic J, Raju R, Naoum C, Knuuti J, Maki M, Underwood RS, Min JK, Elmore K, Stuijfzand WJ, van Royen N, Tulevski II, Somsen AG, Huisman MC, van Lingen AA, Heymans MW, van de Ven PM, van Kuijk C, Lammertsma AA, van Rossum AC, Knaapen P. Comparison of Coronary CT Angiography, SPECT, PET, and Hybrid Imaging for Diagnosis of Ischemic Heart Disease Determined by Fractional Flow Reserve. JAMA Cardiol. 2017 Oct 1;2(10):1100-1107. doi: 10.1001/jamacardio.2017.2471. PMID 28813561
- [Background] Murthy VL, Naya M, Foster CR, Hainer J, Gaber M, Di Carli G, Blankstein R, Dorbala S, Sitek A, Pencina MJ, Di Carli MF. Improved cardiac risk assessment with noninvasive measures of coronary flow reserve. Circulation. 2011 Nov 15;124(20):2215-24. doi: 10.1161/CIRCULATIONAHA.111.050427. Epub 2011 Oct 17. PMID 22007073
- [Background] Dorbala S, Di Carli MF. Cardiac PET perfusion: prognosis, risk stratification, and clinical management. Semin Nucl Med. 2014 Sep;44(5):344-57. doi: 10.1053/j.semnuclmed.2014.05.003. PMID 25234079
- [Background] Taqueti VR, Hachamovitch R, Murthy VL, Naya M, Foster CR, Hainer J, Dorbala S, Blankstein R, Di Carli MF. Global coronary flow reserve is associated with adverse cardiovascular events independently of luminal angiographic severity and modifies the effect of early revascularization. Circulation. 2015 Jan 6;131(1):19-27. doi: 10.1161/CIRCULATIONAHA.114.011939. Epub 2014 Nov 16. PMID 25400060
- [Background] Gould KL, Johnson NP, Bateman TM, Beanlands RS, Bengel FM, Bober R, Camici PG, Cerqueira MD, Chow BJW, Di Carli MF, Dorbala S, Gewirtz H, Gropler RJ, Kaufmann PA, Knaapen P, Knuuti J, Merhige ME, Rentrop KP, Ruddy TD, Schelbert HR, Schindler TH, Schwaiger M, Sdringola S, Vitarello J, Williams KA Sr, Gordon D, Dilsizian V, Narula J. Anatomic versus physiologic assessment of coronary artery disease. Role of coronary flow reserve, fractional flow reserve, and positron emission tomography imaging in revascularization decision-making. J Am Coll Cardiol. 2013 Oct 29;62(18):1639-1653. doi: 10.1016/j.jacc.2013.07.076. Epub 2013 Aug 28. PMID 23954338
- [Background] Taqueti VR, Shaw LJ, Cook NR, Murthy VL, Shah NR, Foster CR, Hainer J, Blankstein R, Dorbala S, Di Carli MF. Excess Cardiovascular Risk in Women Relative to Men Referred for Coronary Angiography Is Associated With Severely Impaired Coronary Flow Reserve, Not Obstructive Disease. Circulation. 2017 Feb 7;135(6):566-577. doi: 10.1161/CIRCULATIONAHA.116.023266. Epub 2016 Nov 14. PMID 27881570
- [Background] Shah NR, Charytan DM, Murthy VL, Skali Lami H, Veeranna V, Cheezum MK, Taqueti VR, Kato T, Foster CR, Hainer J, Gaber M, Klein J, Dorbala S, Blankstein R, Di Carli MF. Prognostic Value of Coronary Flow Reserve in Patients with Dialysis-Dependent ESRD. J Am Soc Nephrol. 2016 Jun;27(6):1823-9. doi: 10.1681/ASN.2015030301. Epub 2015 Oct 12. PMID 26459635
- [Background] Murthy VL, Naya M, Taqueti VR, Foster CR, Gaber M, Hainer J, Dorbala S, Blankstein R, Rimoldi O, Camici PG, Di Carli MF. Effects of sex on coronary microvascular dysfunction and cardiac outcomes. Circulation. 2014 Jun 17;129(24):2518-27. doi: 10.1161/CIRCULATIONAHA.113.008507. Epub 2014 Apr 30. PMID 24787469
- [Background] Murthy VL, Naya M, Foster CR, Gaber M, Hainer J, Klein J, Dorbala S, Blankstein R, Di Carli MF. Association between coronary vascular dysfunction and cardiac mortality in patients with and without diabetes mellitus. Circulation. 2012 Oct 9;126(15):1858-68. doi: 10.1161/CIRCULATIONAHA.112.120402. Epub 2012 Aug 23. PMID 22919001
- [Background] Driessen RS, Danad I, Stuijfzand WJ, Schumacher SP, Knuuti J, Maki M, Lammertsma AA, van Rossum AC, van Royen N, Raijmakers PG, Knaapen P. Impact of Revascularization on Absolute Myocardial Blood Flow as Assessed by Serial [15O]H2O Positron Emission Tomography Imaging: A Comparison With Fractional Flow Reserve. Circ Cardiovasc Imaging. 2018 May;11(5):e007417. doi: 10.1161/CIRCIMAGING.117.007417. PMID 29703779
- [Background] Holubkov R, Laskey WK, Haviland A, Slater JC, Bourassa MG, Vlachos HA, Cohen HA, Williams DO, Kelsey SF, Detre KM; NHLBI Dynamic Registry. Registry Investigators. Angina 1 year after percutaneous coronary intervention: a report from the NHLBI Dynamic Registry. Am Heart J. 2002 Nov;144(5):826-33. doi: 10.1067/mhj.2002.125505. PMID 12422151
- [Background] Arnold SV, Jang JS, Tang F, Graham G, Cohen DJ, Spertus JA. Prediction of residual angina after percutaneous coronary intervention. Eur Heart J Qual Care Clin Outcomes. 2015 Jul 1;1(1):23-30. doi: 10.1093/ehjqcco/qcv010. PMID 29474572
- [Background] Weintraub WS, Spertus JA, Kolm P, Maron DJ, Zhang Z, Jurkovitz C, Zhang W, Hartigan PM, Lewis C, Veledar E, Bowen J, Dunbar SB, Deaton C, Kaufman S, O'Rourke RA, Goeree R, Barnett PG, Teo KK, Boden WE; COURAGE Trial Research Group; Mancini GB. Effect of PCI on quality of life in patients with stable coronary disease. N Engl J Med. 2008 Aug 14;359(7):677-87. doi: 10.1056/NEJMoa072771. PMID 18703470
- [Background] Sdringola S, Gould KL, Zamarka LG, McLain R, Garner J. A 6 month randomized, double blind, placebo controlled, multi-center trial of high dose atorvastatin on myocardial perfusion abnormalities by positron emission tomography in coronary artery disease. Am Heart J. 2008 Feb;155(2):245-53. doi: 10.1016/j.ahj.2007.10.025. Epub 2007 Dec 19. PMID 18215593
- [Background] Gould KL, Ornish D, Scherwitz L, Brown S, Edens RP, Hess MJ, Mullani N, Bolomey L, Dobbs F, Armstrong WT, et al. Changes in myocardial perfusion abnormalities by positron emission tomography after long-term, intense risk factor modification. JAMA. 1995 Sep 20;274(11):894-901. doi: 10.1001/jama.1995.03530110056036. PMID 7674504
- [Background] Gould KL, Martucci JP, Goldberg DI, Hess MJ, Edens RP, Latifi R, Dudrick SJ. Short-term cholesterol lowering decreases size and severity of perfusion abnormalities by positron emission tomography after dipyridamole in patients with coronary artery disease. A potential noninvasive marker of healing coronary endothelium. Circulation. 1994 Apr;89(4):1530-8. doi: 10.1161/01.cir.89.4.1530. PMID 8149518
- [Background] Wielepp P, Baller D, Gleichmann U, Pulawski E, Horstkotte D, Burchert W. Beneficial effects of atorvastatin on myocardial regions with initially low vasodilatory capacity at various stages of coronary artery disease. Eur J Nucl Med Mol Imaging. 2005 Dec;32(12):1371-7. doi: 10.1007/s00259-005-1828-6. Epub 2005 Aug 31. PMID 16133398
- [Background] Schindler TH, Zhang XL, Vincenti G, Mhiri L, Lerch R, Schelbert HR. Role of PET in the evaluation and understanding of coronary physiology. J Nucl Cardiol. 2007 Jul;14(4):589-603. doi: 10.1016/j.nuclcard.2007.05.006. No abstract available. PMID 17679069
- [Background] Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Prodzinski J, McDonell M, Fihn SD. Development and evaluation of the Seattle Angina Questionnaire: a new functional status measure for coronary artery disease. J Am Coll Cardiol. 1995 Feb;25(2):333-41. doi: 10.1016/0735-1097(94)00397-9. PMID 7829785
- [Background] Chan PS, Jones PG, Arnold SA, Spertus JA. Development and validation of a short version of the Seattle angina questionnaire. Circ Cardiovasc Qual Outcomes. 2014 Sep;7(5):640-7. doi: 10.1161/CIRCOUTCOMES.114.000967. Epub 2014 Sep 2. PMID 25185249
- [Background] Rumsfeld JS, Alexander KP, Goff DC Jr, Graham MM, Ho PM, Masoudi FA, Moser DK, Roger VL, Slaughter MS, Smolderen KG, Spertus JA, Sullivan MD, Treat-Jacobson D, Zerwic JJ; American Heart Association Council on Quality of Care and Outcomes Research, Council on Cardiovascular and Stroke Nursing, Council on Epidemiology and Prevention, Council on Peripheral Vascular Disease, and Stroke Council. Cardiovascular health: the importance of measuring patient-reported health status: a scientific statement from the American Heart Association. Circulation. 2013 Jun 4;127(22):2233-49. doi: 10.1161/CIR.0b013e3182949a2e. Epub 2013 May 6. No abstract available. PMID 23648778
- [Background] Spertus JA, Jones P, McDonell M, Fan V, Fihn SD. Health status predicts long-term outcome in outpatients with coronary disease. Circulation. 2002 Jul 2;106(1):43-9. doi: 10.1161/01.cir.0000020688.24874.90. PMID 12093768
- [Background] McNamara RL, Spatz ES, Kelley TA, Stowell CJ, Beltrame J, Heidenreich P, Tresserras R, Jernberg T, Chua T, Morgan L, Panigrahi B, Rosas Ruiz A, Rumsfeld JS, Sadwin L, Schoeberl M, Shahian D, Weston C, Yeh R, Lewin J. Standardized Outcome Measurement for Patients With Coronary Artery Disease: Consensus From the International Consortium for Health Outcomes Measurement (ICHOM). J Am Heart Assoc. 2015 May 19;4(5):e001767. doi: 10.1161/JAHA.115.001767. PMID 25991011
- [Background] Rose GA, Blackburn H. Cardiovascular survey methods. Monogr Ser World Health Organ. 1968;56:1-188. No abstract available. PMID 4972212
- See also: Reference #30 — https://www.cms.gov/Medicare/Quality-Initiatives-Patient-Assessment-Instruments/MMS/Downloads/Hospital-Level-PRO-Based-PM-for-Patients-Undergoing-non-Emergent-PCI_Public-Comment-Summary-Report.pdf